CLINICAL TRIAL: NCT03538275
Title: Chronobiology and Depression: Circadian Analytics as a Biomarker for Diagnosis and Longitudinal Monitoring of Depressive Subtypes
Brief Title: Chronobiology and Depression: Circadian Analytics as a Biomarker for Depressive Subtypes
Status: Completed | Type: Observational
Sponsor: Medibio Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: MB-DEPMON01
Record Dates: First submitted 2018-05-03; First posted 2018-05-29 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Depression, Bipolar; Depression, Unipolar; Healthy
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Unipolar depression cohort: Subjects with a known Dx of unipolar depression.
  Interventions: Other: Monitoring test
- Bipolar depression cohort: Subjects with a known Dx of bipolar disorder
  Interventions: Other: Monitoring test
- Healthy Control cohort: Subjects with no known unipolar or bipolar Dx.
  Interventions: Other: Monitoring test

INTERVENTIONS:
Other: Monitoring test — Participants wear Zephyr BioPatch for three 24-hour periods and ZMachine Insight for three sleep periods.

SUMMARY:
An objective measure of treatment response could be a valuable new tool in the armamentarium of depression management, and this holds true for stimulation-based and pharmacological therapies alike. Hence, the Medibio Depression Monitoring Study will use the Medibio analytics platform to characterize autonomic, circadian, and sleep patterns before and during the initial 8 weeks of pharmacologic therapy for moderate-to-severe depression. The study will also explore any differences in these measures between treatment responders and non-responders, and between depression subtypes, including bipolar and unipolar depression. The study will also characterize longitudinal, ambulatory EEG measures throughout the observation period.

DETAILED DESCRIPTION:
This longitudinal, two-phase, three-arm, exploratory, observational study will use the Medibio analytics platform-with heart rate, activity, postural, and EEG data inputs-to characterize autonomic, circadian, and sleep patterns in unipolar depressed and bipolar depressed patients, which will include those with atypical and melancholic subtypes, undergoing the initial phase of standard pharmacological treatment, as well as in a non-depressed control group.

Phase I will serve as a non-blinded, discovery phase for Medibio algorithm development.

Phase II is optional, based upon sponsor/investigator assessment of results from Phase I. Phase II procedures will be identical to those in Phase I, with the exception that the Medibio algorithm will be blinded to clinical classification and status.

The study cohorts will comprise: a) individuals initiating standard pharmacologic therapy with SSRIs for moderate-to- severe unipolar depression (will include subjects with melancholic and atypical subtypes), b) individuals initiating standard pharmacologic therapy with lamotrigine, lithium, or valproate for moderate or severe bipolar I or II depression (will also include subjects with melancholic and atypical subtypes), and c) non-depressed individuals who have been matched at the group level for age and gender (control subjects). Before the commencement of pharmacologic therapy (Baseline, t=0), at t=4 weeks, and at t=8 weeks, heart rate, activity, postural data will be collected using the Zephyr BioPatch (Medtronic, Inc.) and ambulatory EEG data will be collected using the ZMachine Insight (General Sleep Corp). Recordings at each time point will consist of three 24-hour Zephyr recordings and three overnight ZMachine recordings.

Clinical assessments will also be captured at the same time points, comprising both clinician-administered instruments [Clinical Global Impression (CGI), Hamilton Depression Rating Scale-17 (HAMD-17), and Young Mania Rating Scale (YMRS)] and subject self-rated instruments [Patient Health Questionnaire-9 (PHQ-9) and Quick Inventory of Depressive Symptomatology-Self Report (QIDS SR16)]. Zephyr and ZMachine data will be filtered based on quality (duration and completeness) and may be 'de-noised,' then will be processed by the Medibio platform to generate autonomic, circadian, and sleep metrics for use in the statistical analysis of study results.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide consent.
* Subject has ability to read and understand the instructions for the study.
* Subject is willing to adhere to study procedures.

Exclusion Criteria:

1. Subject has presence of mild, moderate, or severe Major Depressive Disorder Episode, based on DSM-IV criteria for diagnosis as documented by clinician administered M.I.N.I OR HAMD-17 rating scale score >7.
2. Subject has bipolar disorder.
3. Subject has active psychotic symptoms.
4. Subject has known or is suspected to have a personality disorder.
5. Subject has current suicidality of medium or high risk as determined by M.I.N.I. or HAMD-17 item #3 score of 3 of higher.
6. Subject has history of central or obstructive sleep apnea OR has a STOP-BANG score of ≥5 OR has a Home Sleep Test assessment (ApneaLink, ResMed) demonstrating AHI≥15.
7. Subject has a pacemaker.
8. Subject currently uses benzodiazepines, sedative-hypnotics, or trazadone on a scheduled basis OR will be likely be prescribed such medication during the 8-week observational phase of the study.
9. Subject currently uses antipsychotic medication for any indication OR will be likely be prescribed such medication during the 8-week observational phase of the study.
10. Subject currently uses chronotropic medication, such as beta-blockers, digoxin, sinoatrial/atrioventricular nodal-acting calcium channel blockers, and amiodarone.
11. Subject is suspected or known to have active alcohol or drug abuse (including but not limited to abuse of marijuana).
12. Subject has a terminal illness.
13. For female subjects, subject is currently known to be pregnant or lactating.
14. Subject has any other acute or chronic condition that in the investigators opinion would preclude the subject from being able to meet all of the protocol requirements, or would compromise the subject's safety during participation in the study, as judged by the investigator.
15. Subject is currently participating in another clinical study, or participated in a clinical study in the past 30 days during which an investigational device or drug was used.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled at 1 site in the United States. Depressed subjects (bipolar and unipolar sub-types) will be recruited from outpatient clinics via direct physician referral and flyers. The study should be conducted with adequate representation of men and women; a minimum enrollment of 25% male subjects is desired. There are no enrollment restrictions based upon race or ethnic origin.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Medibio platform classification | Through study completion, an average of 8 weeks
  The Medibio platform will use 24 hours recording to monitor disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Bruner, Study Director — Medibio Limited
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided